CLINICAL TRIAL: NCT01047384
Title: Management of Postoperative Pain Following Total Knee Arthroplasty by Using Acupuncture-moxibustion Therapy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: acupuncture
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2010-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Experimental (Experimental): acupuncture-moxibustion therapy
  Interventions: Procedure: acupuncture-moxibustion therapy
- Regular therapy (Active Comparator): Regular therapy
  Interventions: Procedure: Regular therapy

INTERVENTIONS:
Procedure: acupuncture-moxibustion therapy
  Arms: Experimental
Procedure: Regular therapy
  Arms: Regular therapy

SUMMARY:
Orthopedic surgery is reportedly among the most painful surgical procedures. Surgical damage following major orthopedic surgery often involves a large, deep incision with considerable tissue dissection and muscle, bone, and vascular exposure. Post-operative pain after such surgery is exacerbated on movement or by reflex spasms of the muscles, which may delay mobilization, reduce satisfaction, prolong hospitalization, and possibly increase medical costs.

We design a prospective randomized study for postoperative pain control following total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for surgery of osteoarthritis of knee
* ability to tolerate surgery under general anesthesia.

Exclusion Criteria:

* refusal or the lack of mental ability to provide informed consent
* neuropathic pain or sensory disorders in the leg requiring surgery
* previous surgery of the knee joint
* coagulation abnormalities
* chronic opioid users
* known history of intolerance to acupuncture-moxibustion therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pain VAS score | pre-operaton, immediately post operation, postop 6hrs, postop 12hrs, postop 18hrs, postop 24hrs, post op 48hrs, postop 72hrs

SECONDARY OUTCOMES:
Functional score: SF-36 | Pre-operation, immediately post-operation, postop 6 weeks, postop 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kweishian, Taoyuan, Taiwan